CLINICAL TRIAL: NCT05778734
Title: StuDy AimED at Increasing AlCohol AbsTinEnce (DEDICATE)
Brief Title: StuDy AimED at Increasing AlCohol AbsTinEnce
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Hagar Hallihan, Postdoctoral Research Fellow, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-1047
Record Dates: First submitted 2023-02-27; First posted 2023-03-21 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: K99 Phase is a single arm study, whiles the R00 phase is a 2-arm study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Other): For the R00 phase: CM-PST treatment group will receive CM-PST intervention, which will consist of 8 sessions total, delivered remotely via Zoom videoconferences in individual sessions over 12 weeks. The first 4 sessions will be delivered weekly, and the remaining 4 sessions every other week. CM-PST will teach participants problem-solving skills using a structured 5-step method. In addition, participants will receive incentives for alcohol abstinence and submission of urine samples twice/wk.
  K99 phase participants will also receive CM-PST intervention.
  Interventions: Behavioral: CM-PST
- Control group (Other): For the R00 phase: Participants in CM-only control will receive incentives for alcohol abstinence and submission of urine samples twice/wk. Participant incentives will start at a $10 gift card, with a $5 increase each subsequent measurement point on which alcohol is not detected or reported, to a maximum of $25, but no gift card on days when alcohol use is detected or reported, and the gift card reinforcer value will be re-set to $10.
  Interventions: Behavioral: CM only

INTERVENTIONS:
Behavioral: CM-PST — CM-PST is a tailored behavioral intervention that enables young adults with AUD to successfully manage and overcome everyday life challenges influencing their alcohol intake.
  Arms: Treatment group
Behavioral: CM only — CM is a behavior therapy that rewards individuals for evidence of positive change (alcohol abstinence).
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to test the feasibility & acceptability of an integrated CM-PST intervention (in K99 phase) and preliminary efficacy (in R00 phase), vs. CM alone, to improve treatment efficacy and inform about neural mechanisms of treatment effects in young adults with Alcohol Use Disorder (AUD).

The aims are as follows:

K99 Aim: Test feasibility & acceptability of a developed CM-PST, by meeting these benchmarks: 2a Feasibility: enroll 20 participants in the new CM-PST in a single-arm pre- and post-study, and retain ≥85% at wk 12. 2b Deliver CM-PST at ≥90% fidelity to intervention protocol. 2c Acceptability to participants: Achieve mean score ≥3 on Client Satisfaction Scale Questionnaire and satisfaction from semi-structured interviews.

R00 Aim 1) Test preliminary efficacy of CM-PST in a 2-arm pilot RCT: Male/female young adults (aged18-24) who meet AUD criteria will be randomized to CM-PST or CM-only control, and assessed at baseline (0), 3, and 6 months. Primary study endpoint will be 3 months.

R00 Aim 2 (Exploratory) Explore potential neural mechanisms of CM-PST effects, by fMRI scanning & analyses of core regions of the brain circuits regulating positive affect (ventral striatum), negative affect (amygdala), and cognitive control (dorsolateral prefrontal cortex), and connectivity between these core regions.

DETAILED DESCRIPTION:
Study Design Formative (K99 Phase), we will test feasibility & acceptability of integrated CM-PST. To test CM-PST, we will recruit/enroll 20 participants in a single-arm pre/post study. Participants who meet eligibility will be invited to our clinical lab at UIC for informed consent and baseline measures. Consenting participants will receive CM-PST intervention via videoconferences such as zoom, in 8 CM-PST individual sessions, every week for sessions 1-4 and every other week for sessions 5-8, over 12 weeks. Participants will complete the Client Satisfaction Scale survey after each session and 3 mo. post-intervention, to quantify their overall experiences with this new CM-PST.

Preliminary efficacy trial (R00 Phase). This will be a 2-arm Randomized control trial in young adults aged 18-24 yr who meet AUD criteria. Prospective participants who respond to our advertisements will be screened by phone for eligibility and to determine their AUD diagnostic status and severity (mild, moderate, severe). Participants who meet eligibility will be invited to our UIC clinical lab for informed consent, baseline self-report measures, urine alcohol screening, and baseline fMRI, and then randomized to either CM-PST (42 participants) or CM-only (42 participants) control group. All participants will complete follow-up assessments at 3 & 6 months with blinded outcome assessors.

ELIGIBILITY:
Inclusion Criteria:

* Male and female young adults aged 18-24 yr
* English-speaking
* Current alcohol use greater or equal to 1 day/week via phone screening, and meet criteria for (past year) mild, moderate or severe AUD on the AUDIT and AUDADIS surveys.
* Completion of written informed consent
* Baseline screening study visit.

Exclusion Criteria:

* Participation in past 6 mo. in AUD or substance use treatment
* Current use of medications used to treat AUD (e.g., naltrexone)
* Lifetime DSM-5 diagnosis of schizophrenia, bipolar disorder, or any psychotic disorder.
* Current use of psychoactive drugs, determined by positive drug toxicology screen
* Conditions (e.g., tic disorder) that would interfere with psychophysiological indices of reward functioning
* Pregnancy or intention to become pregnant
* Additional exclusion criteria pertaining to fMRI scan in R00 phase only: a) bodily ferrous metals (e.g., aneurysm clips, shrapnel/retained particles) or b) claustrophobia, inability to tolerate small enclosed spaces.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2023-07-30 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Alcohol abstinence. | Up to 6months
  Participants will be monitored for 6 months to assess alcohol abstinence by blood alcohol content.

SECONDARY OUTCOMES:
Change in AUD severity at 3 months. | Baseline, 3months.
  Measured by Alcohol Use Disorder and Associated Disabilities Interview Schedule-5. Change in AUD severity from baseline to 3 months.
Change in AUD severity at 6 months. | Baseline, 6months.
  Measured by Alcohol Use Disorder and Associated Disabilities Interview Schedule-5. Change in AUD severity from baseline to 6 months.
Change in AUD screening status. | Up to 6months.
  Measured by AUDIT. Participants will be monitored for up to 6 months. This is the number of participants who screen positive for AUD.
Change in Alcohol-related negative consequences at 3 months. | Baseline, 3 months.
  Measured by Rutgers Alcohol Problem Index (RAPI).
Change in Alcohol-related negative consequences at 6 months. | Baseline, 6 months.
  Measured by Rutgers Alcohol Problem Index (RAPI).
Change in Alcohol use at 3 months. | Baseline, 3 months.
  Measured by 90-day Timeline Followback (TLFB).
Change in Alcohol use at 6 months. | Baseline, 6 months.
  Measured by 90-day Timeline Followback (TLFB).
Change in Drug use at 3 months. | Baseline, 3 months.
  Measured by 90-day Timeline Followback (TLFB).
Change in Drug use at 6 months. | Baseline, 6 months.
  Measured by 90-day Timeline Followback (TLFB).
Change in Reasons for drinking at 3 months. | Baseline, 3 months
  Measured by Drinking Motives Questionnaire Revised (DMQ-R).
Change in Reasons for drinking at 6 months. | Baseline, 6 months
  Measured by Drinking Motives Questionnaire Revised (DMQ-R).
Change in negative affect at 3 months. | Baseline, 3 months
  Measured by Positive and Negative Affect Schedule (PANAS).
Change in negative affect at 6 months. | Baseline, 6 months
  Measured by Positive and Negative Affect Schedule (PANAS).
Change in positive affect at 3 months. | Baseline, 3 months
  Measured by Positive and Negative Affect Schedule (PANAS).
Change in positive affect at 6 months. | Baseline, 6 months
  Measured by Positive and Negative Affect Schedule (PANAS).
Change in Neural target engagement of positive affect. affect (ventral striatum), negative affect (amygdala), and cognitive control (dorsolateral prefrontal cortex). | Baseline, 3 months.
  Measured by Functional magnetic resonance imaging (fMRI).

OTHER OUTCOMES:
Intervention Acceptability (K99 phase only). | 3 months
  Measured by Client Satisfaction Questionnaire.
Intervention Acceptability from interviews (K99 phase only). | 3 months
  Measured by satisfaction from semi-structured interviews.
Intervention Fidelity (K99 phase only). | 3 months
  Participant adherence to the CM-PST intervention schedule will be assessed by documented session attendance.
Participant Retention (K99 phase only). | Up to 6 months.
  Participant retention will be assessed throughout the study by monitoring the proportion of the sample retained at 3-months and 6-months.

CONTACTS AND LOCATIONS:
Overall Officials: Hagar Hallihan, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
We will adhere to the NIH Grant Policy on Sharing of Unique Research Resources including the Principles and Guidelines for Recipients of NIH Research Grants and Contracts on Obtaining and Disseminating Biomedical Research Resources issued December 23, 1999. Data from this research will be shared and the results of this research will be made available via publication in scientific journals and through scientific meetings where our findings are reported. Publication of data shall occur during the project, if appropriate, or at the end of the project, consistent with typical scientific practices. All publications will be made publicly available consistent with NIH policies.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After analyzing.

REFERENCES:
- [Derived] Hallihan H, Lee S, Rospenda KM, Wu Y, Adomah R, Knepper A, Ma J. Feasibility and acceptability of contingency management and problem-solving therapy intervention for enhancing alcohol abstinence: a single-arm, mixed methods pilot clinical trial. BMJ Open. 2025 Aug 19;15(8):e098691. doi: 10.1136/bmjopen-2024-098691. PMID 40829841